CLINICAL TRIAL: NCT04591223
Title: Testing the Competency-based Theory of Change for Suicide Risk Among Young Male Internet Users With Societal Masculinity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr.Yik-Wa Law, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17602620
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Self-Harm, Deliberate; Suicidal Ideation; Masculinity
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Masculinity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + six weekly sessions of competency-based module (CbM) (Experimental): This group of participants will be receiving online social work (OSW) treatment as usual (TAU) from NGO service provider as well as a well-designed, one on one structural physical workout module to be offered by a licensed senior physical trainer in public sports ground or gymnasium.
  Interventions: Behavioral: Competency-based physical training (CbM)
- TAU (No Intervention): This group of participants will be receiving online social work (OSW) treatment as usual (TAU) from NGO service provider.

INTERVENTIONS:
Behavioral: Competency-based physical training (CbM) — The intervention to be added to online social work treatment as usual (OSW) is a well-designed, one-on-one structural physical workout module which will be offered by a licensed senior physical trainer in public sports ground or gymnasium. The aim is to strengthen participants' sense of competence, improve their physical fitness, self-confidence and self-image through an outcome-driven Circuit training. One of the chief advantages of Circuit training is its adaptability. Circuit training can be performed with gym equipment and/or bodyweight exercises which is deemed to be suitable for beginner and easy to practice at home on oneself. Participants can continue to replicate the exercise with or without any equipment. The program will be delivered in six one-hour sessions, including face-to-face and online mode, over one month.
  Arms: TAU + six weekly sessions of competency-based module (CbM)

SUMMARY:
To propose a competency-based theory of change for reducing suicide risks among male Internet users with salient traits of societal masculinity; To test whether the theory of change using the competency-based model has additional effects on reducing self-harm and/or suicidal ideation in addition to the online social work treatment-as-usual model; To provide online social work service providers with evidence-based measures for reducing the risks of self-harm and/or suicide among young male Internet users.

DETAILED DESCRIPTION:
This is a randomized waitlist-controlled trial of 60 participants examining the effects of a proposed competency-based model on self-harm relative to those of OSW alone. In the online survey (T0), subjects with self-harm or suicidal ideation will be invited to give informed consent, and then be randomly assigned to one of two groups: 1) OSW (control), or 2) OSW + six weekly sessions of competency-based physical training (intervention). They will be assessed at three measurement time points (T1 = one-month; T2 = three-month; and T3 = five-month from T0 at post-intervention). The intervention group is hypothesized to display a greater reduction in the primary outcomes of self-harm and suicidal ideation than the OSW group. Chi-square tests giving p <=0.05 will indicate a goodness of fit of the linear mixed model, which address random effects in the data and handles intention-to-treat (ITT).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who meet the cut-off of 1.0 on the Chinese Adult Suicidal Ideation Questionnaire (ASIQ4); Self-injury incidents in the past 12 months

Exclusion Criteria:

* Individuals with severe physical disabilities

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male Internet user
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Adult Suicidal Ideation at 1-month, 3-month and 5-month | Baseline,1-month, 3-month, 5-month
  Change in scores on Suicidal ideation as measured by the self-report the Adult Suicidal Ideation Questionnaire (ASIQ-4) - the four-item short form in Chinese, scoring on a 7-point scale ranging from 0 to 24.
  A higher score on the scale suggests a higher risk of suicide.
Change from baseline measurement of hopelessness at 1-month, 3-month and 5-month | Baseline, 1-month, 3-month, 5-month
  Hopelessness will be assessed by four questions measuring hopelessness extracted from the Beck Hopelessness Scale (BHS4), scoring on a 6-point scale ranging from 0 to 20.
  A higher score on the scale suggests a higher levels of depression, suicidal intent, and/or ideation.
Change from baseline measurement of depression at 1-month, 3-month and 5-month | Baseline, 1-month, 3-month, 5-month
  Depression will be assessed via 12 questions from the short-form General Health Questionnaire (GHQ-12), scoring on a 4-point scale ranging from 0 to 36.
  A higher score on the scale suggests a higher level of emotional distress and depression.
Change of baseline sense of competency at 1-month, 3-month and 5-month | Baseline, 1-month, 3-month, 5-month
  Sense of competency will be assessed via 40 questions from the Chinese Physical Self-Description Questionnaire-Short Form (CPSDQ-S), scoring on a 6-point scale ranging from 0 to 200.
  A higher score suggest a higher level of self-perceived physical competency and self-esteem.
Change of baseline perceived social support at 1-month, 3-month and 5-month | Baseline, 1-month, 3-month, 5-month
  Social support will be assessed using the Chinese version of the Multidimensional Scale of Perceived Social Support (MSPSS-C). The MSPSS measures the degree of social support received from family, friends, and significant others, and has been proven to have good internal and test-retest reliability and moderate construct validity
Change of baseline measurements of weight (body composition) at 1-month, 3-month, 5-month | Baseline, 1-month, 3-month, 5-month
  Weight, as a one of the indicators of body composition, will be measured in kilograms at four different time points.
Change of baseline measurements of skinfold (body composition) at 1-month, 3-month, 5-month | Baseline, 1-month, 3-month, 5-month
  A skinfold caliper will be used to assess the skinfold thickness, which is considered to be one of the indicators of body composition.
Change of baseline measurements of hip and waist girth (body composition) at 1-month, 3-month, 5-month | Baseline, 1-month, 3-month, 5-month
  Both hip and waist girth will be measured in inches at four different time points as part of the measurement of body composition.
Change of baseline measurement of self-reported compliance to service at baseline, 1-month, 3-month, 5-month | Baseline, 1-month, 3-month, 5-month
  Questionnaire will be distributed to subjects to assess their compliance to service: frequency of service use, including medical and psychosocial services at four different time points.
Change of baseline measurement of suicidal behavior at 1-month, 3-month, 5-month | Baseline, 1-month, 3-month, 5-month
  Subjects were expected to answer three separate questions with dichotomous yes/no responses: in the past few weeks, (1) have you thought about committing suicide? 2) have you been actively planning to commit suicide? 3) did you make any suicide attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Yik Wa Law, Principal Investigator — The University of Hong Kong; Sik-ying Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No